CLINICAL TRIAL: NCT02290340
Title: A Phase 1b/2a Randomized, Double-Blind, Placebo-controlled, Dose-escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of MEDI8897, a Monoclonal Antibody With an Extended Half-life Against Respiratory Syncytial Virus, in Healthy Preterm Infants
Acronym: MEDI8897 1b
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: D5290C00002
Record Dates: First submitted 2014-10-17; First posted 2014-11-14 (Estimated); Results first posted 2018-09-19 (Actual); Last update posted 2018-09-19 (Actual); Status verified 2018-09

CONDITIONS: Respiratory Syncytial Virus
Keywords: Respiratory Syncytial Virus, RSV

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Participants will receive placebo intramuscularly.
  Interventions: Drug: Placebo
- MEDI8897 10 mg (Experimental): Participants will receive a single dose of MEDI8897 10 milligram (mg) intramuscularly.
  Interventions: Drug: MEDI8897 10 mg
- MEDI8897 25 mg (Experimental): Participants will receive a single dose of MEDI8897 25 mg intramuscularly.
  Interventions: Drug: MEDI8897 25 mg
- MEDI8897 50 mg (Experimental): Participants will receive a single dose of MEDI8897 50 mg intramuscularly.
  Interventions: Drug: MEDI8897 50 mg

INTERVENTIONS:
Drug: Placebo — Participants will receive placebo intramuscularly.
  Arms: Placebo
Drug: MEDI8897 10 mg — Participants will receive a single dose of MEDI8897 10 milligram (mg) intramuscularly.
  Arms: MEDI8897 10 mg
Drug: MEDI8897 25 mg — Participants will receive a single dose of MEDI8897 25 mg intramuscularly.
  Arms: MEDI8897 25 mg
Drug: MEDI8897 50 mg — Participants will receive a single dose of MEDI8897 50 mg intramuscularly.
  Arms: MEDI8897 50 mg

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and pharmacokinetics of an extended half-life anti-respiratory syncytial virus (RSV) monoclonal antibody compared to placebo when administered to healthy preterm infants.

DETAILED DESCRIPTION:
This Phase 1b/2a study will be a dose-escalation design to begin data collection on PK and safety in children. The population to be enrolled is healthy preterm infants born between 32 weeks 0 days and 34 weeks 6 days gestation who would not receive RSV prophylaxis based on the American Academy of Pediatrics (AAP) or other local guidelines. These subjects will not be receiving palivizumab, allowing for a placebo comparator group to begin collecting data on incidence rates of RSV medically attended lower respiratory illness (MA-LRI) and efficacy. Enrollment is planned at approximately 20 sites in the USA, Chile, and South Africa.

ELIGIBILITY:
Key Inclusion Criteria:

* Healthy infants born between 32 weeks 0 days and 34 weeks 6 days gestational age
* Infants who are entering their first RSV season at the time of screening

Key Exclusion Criteria:

* Gestational age < 32 weeks 0 days and >34 weeks 6 days
* Meets AAP or other local criteria to receive commercial palivizumab
* Any fever (≥ 100.4°F [≥ 38.0°C], regardless of route) or lower respiratory illness within 7 days prior to randomization
* Acute illness (defined as the presence of moderate or severe signs and symptoms) at the time of randomization
* Active RSV infection (a child with signs/symptoms of respiratory infection must have negative RSV testing) or known prior history of RSV infection
* Receipt of palivizumab or any RSV vaccine, including maternal RSV vaccination

Max Age: 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 151 (Actual)
Dates: Start 2015-01-13 (Actual); Primary Completion 2016-09-28 (Actual); Study Completion 2016-09-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (7):
  - Research Site, Anaheim, California
  - Research Site, Ontario, California
  - Research Site, Syracuse, New York
  - Research Site, Cleveland, Ohio
  - Research Site, Charleston, South Carolina
  - Research Site, St. George, Utah
  - Research Site, Marshfield, Wisconsin
- Chile (2):
  - Research Site, Santiago
  - Research Site, Valdivia
- South Africa (4):
  - Research Site, Cape Town
  - Research Site, East London
  - Research Site, Johannesburg
  - Research Site, Pretoria

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between January 2015 and September 2015 at 10 sites (USA, South Africa, and Chile) and followed for 1 year after dosing.
Pre-assignment Details: A total of 151 participants were screened in the study, of which 89 participants were randomized and treated.
Groups:
- Placebo: Participants received placebo intramuscularly.
- MEDI8897 10 mg: Participants received a single dose of MEDI8897 10 milligram (mg) intramuscularly.
- MEDI8897 25 mg: Participants received a single dose of MEDI8897 25 mg intramuscularly.
- MEDI8897 50 mg: Participants received a single dose of MEDI8897 50 mg intramuscularly.
Period: Overall Study
Arm/Group | Placebo | MEDI8897 10 mg | MEDI8897 25 mg | MEDI8897 50 mg
Started | 18 | 8 | 31 | 32
Completed | 16 | 8 | 31 | 30
Not Completed | 2 | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Not completed — Other | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The As-treated Population included all participants who received any study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | MEDI8897 10 mg | MEDI8897 25 mg | MEDI8897 50 mg | Total
Number analyzed (Participants) | 18 | 8 | 31 | 32 | 89
Age, Continuous [Mean (Standard Deviation); unit: Months] | 7.0 (2.6) | 4.2 (2.1) | 6.7 (2.7) | 6.9 (2.5) | 6.6 (2.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 4 | 19 | 19 | 53
  Male | 7 | 4 | 12 | 13 | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 10 | 1 | 19 | 21 | 51
  White | 4 | 6 | 0 | 2 | 12
  More than one race | 0 | 1 | 0 | 1 | 2
  Unknown or Not Reported | 4 | 0 | 11 | 7 | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) is any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening situation (immediate risk of dying); persistent or significant disability/incapacity of a participant who received MEDI8897. TEAEs and TESAEs were the events that occurred between administration of study drug (Day 1) and Day 361 that were absent before treatment or that worsened relative to pre-treatment state.
Time Frame: From Study Drug Administration (Day 1) Through the Follow-up Period (Day 361)
Population: The As-treated Population included all participants who received any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI8897 10 mg | MEDI8897 25 mg | MEDI8897 50 mg
Number analyzed (Participants) | 18 | 8 | 31 | 32
Participants
  TEAEs | 17 | 5 | 31 | 30
  TESAEs | 0 | 0 | 1 | 2

2. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events of Special Interest
Description: An AESI was one of scientific and medical interest specific to understanding of study product and may have required close monitoring and rapid communication by investigator (that is, within 24 hrs of knowledge of the event) to the sponsor. The AESIs for this study were hepatic function abnormality meeting the definition of Hy's law, hypersensitivity reactions including anaphylaxis, immune complex disease, and thrombocytopenia. Treatment-emergent AESIs were collected from the time of dosing until Day 361 post-dose.
Time Frame: From Study Drug Administration (Day 1) Through the Follow-up Period (Day 361)
Population: The As-treated Population included all participants who received any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI8897 10 mg | MEDI8897 25 mg | MEDI8897 50 mg
Number analyzed (Participants) | 18 | 8 | 31 | 32
Participants | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Clinical Laboratory Abnormalities Reported as Treatment-Emergent Adverse Events
Description: Laboratory abnormalities determined by the investigator to be clinically significant that occurred after study drug dosing through 151 days post-dose that were absent before treatment or that worsened relative to pre-treatment state were reported as TEAEs. Laboratory evaluations (haematology and serum chemistry) of blood samples were performed.
Time Frame: From Study Drug Administration (Day 1) Through the Follow-up Period (Day 151)
Population: The As-treated Population included all participants who received any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI8897 10 mg | MEDI8897 25 mg | MEDI8897 50 mg
Number analyzed (Participants) | 18 | 8 | 31 | 32
Participants
  Anaemia | 6 | 0 | 8 | 4
  Microcytic anaemia | 0 | 0 | 0 | 3
  Neutropenia | 0 | 0 | 0 | 1

4. Secondary Outcome: Time to Reach Maximum Observed Serum Concentration (Tmax) of MEDI8897
Description: The Tmax defined as time at which maximum observed concentration of MEDI8897 (Cmax) was observed.
Time Frame: Pre-dose at Baseline (Days -7 to -1) and on Days 7 (± 1), 30 (± 5), 150 (± 7) and 360 (± 7) Post-dose
Population: The As-treated Population included all participants who received any study drug. Here, "N" signifies number of participants analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: Day
Arm/Group | MEDI8897 10 mg | MEDI8897 25 mg | MEDI8897 50 mg
Number analyzed (Participants) | 5 | 29 | 31
Day | 7.04 (0.0683) | 7.04 (0.394) | 6.93 (0.549)

5. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of MEDI8897
Description: The Cmax is the maximum observed serum concentration of MEDI8897.
Time Frame: Pre-dose at Baseline (Days -7 to -1) and on Days 7 (± 1), 30 (± 5), 150 (± 7) and 360 (± 7) Post-dose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: microgram per milliliter (mcg/mL)
Arm/Group | MEDI8897 10 mg | MEDI8897 25 mg | MEDI8897 50 mg
Number analyzed (Participants) | 5 | 29 | 31
microgram per milliliter (mcg/mL) | 23.2 (9.28) | 30.9 (10.4) | 71.7 (15.9)

6. Secondary Outcome: Area Under the Concentration-Time Curve From Day 1 to Day 151 (AUC [1-151]) of MEDI8897
Description: Area under the concentration-time curve of the MEDI8897 in serum over the time interval from day 1 to day 151 (AUC1-151).
Time Frame: Pre-dose at Baseline (Days -7 to -1) and on Days 7 (± 1), 30 (± 5), and 150 (± 7) Post-dose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Day*mcg/mL
Arm/Group | MEDI8897 10 mg | MEDI8897 25 mg | MEDI8897 50 mg
Number analyzed (Participants) | 5 | 29 | 31
Day*mcg/mL | 1940 (809) | 2260 (881) | 5470 (1440)

7. Secondary Outcome: Area Under the Concentration-Time Curve From Zero to Infinity (AUC [0-infinity]) of MEDI8897
Description: The pharmacokinetic (PK) parameter AUC (0-infinity) was estimated based on the serum concentrations of MEDI8897.
Time Frame: Pre-dose at Baseline (Days -7 to -1) and on Days 7 (± 1), 30 (± 5), 150 (± 7) and 360 (± 7) Post-dose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Day*mcg/mL
Arm/Group | MEDI8897 10 mg | MEDI8897 25 mg | MEDI8897 50 mg
Number analyzed (Participants) | 1 | 6 | 14
Day*mcg/mL | 2450 (NA) — Standard Deviation was not evaluable due to insufficient numbers of participants. | 4320 (1070) | 7510 (1870)

8. Secondary Outcome: Terminal Elimination Half Life (t1/2) of MEDI8897
Description: Terminal phase elimination half-life (t1/2) is the time required for half of the drug to be eliminated from the serum.
Time Frame: Pre-dose at Baseline (Days -7 to -1) and on Days 7 (± 1), 30 (± 5), 150 (± 7) and 360 (± 7) Post-dose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Day
Arm/Group | MEDI8897 10 mg | MEDI8897 25 mg | MEDI8897 50 mg
Number analyzed (Participants) | 1 | 6 | 14
Day | 72.9 (NA) — Standard Deviation was not evaluable due to insufficient numbers of participants. | 66.2 (7.83) | 62.5 (9.35)

9. Secondary Outcome: Extravascular Clearance (CL/F) of MEDI8897
Description: Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the body.
Time Frame: Pre-dose at Baseline (Days -7 to -1) and on Days 7 (± 1), 30 (± 5), 150 (± 7) and 360 (± 7) Post-dose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mL/day
Arm/Group | MEDI8897 10 mg | MEDI8897 25 mg | MEDI8897 50 mg
Number analyzed (Participants) | 1 | 6 | 14
mL/day | 4.08 (NA) — Standard Deviation was not evaluable due to insufficient numbers of participants. | 6.05 (1.31) | 7.01 (1.57)

10. Secondary Outcome: Extravascular Volume of Distribution (Vz/F) of MEDI8897
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired serum concentration of a drug.
Time Frame: Pre-dose at Baseline (Days -7 to -1) and on Days 7 (± 1), 30 (± 5), 150 (± 7) and 360 (± 7) Post-dose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | MEDI8897 10 mg | MEDI8897 25 mg | MEDI8897 50 mg
Number analyzed (Participants) | 1 | 6 | 14
mL | 429 (NA) — Standard Deviation was not evaluable due to insufficient numbers of participants. | 581 (159) | 633 (168)

11. Secondary Outcome: Number of Participants Positive for Anti-Drug Antibodies to MEDI8897
Description: A participant was considered ADA-positive if the participant had a positive reading at any time point post baseline. Titers greater than or equal to 50 were considered positive.
Time Frame: Pre-dose at Baseline (Days -7 to -1) and on Days 31, 151, and 361 Post-dose
Population: The As-treated Population included participants who received any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI8897 10 mg | MEDI8897 25 mg | MEDI8897 50 mg
Number analyzed (Participants) | 18 | 8 | 31 | 32
Participants
  Baseline | 1 | 0 | 0 | 0
  Day 31: number analyzed (Participants) | 16 | 5 | 29 | 32
  Day 31 | 0 | 2 | 0 | 0
  Day 151: number analyzed (Participants) | 14 | 6 | 31 | 32
  Day 151 | 0 | 0 | 0 | 0
  Day 361: number analyzed (Participants) | 16 | 8 | 31 | 29
  Day 361 | 0 | 1 | 7 | 10

ADVERSE EVENTS:
Time Frame: From Study Drug Administration (Day 1) Through the Follow-up Period (Day 361)
Arm/Group | Placebo | MEDI8897 10 mg | MEDI8897 25 mg | MEDI8897 50 mg
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/8 | 0/31 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/8 | 1/31 | 2/32
Other Adverse Events (participants affected / at risk) | 17/18 | 5/8 | 31/31 | 28/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=18) | MEDI8897 10 mg (N=8) | MEDI8897 25 mg (N=31) | MEDI8897 50 mg (N=32)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Febrile convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=18) | MEDI8897 10 mg (N=8) | MEDI8897 25 mg (N=31) | MEDI8897 50 mg (N=32)
Anaemia (Blood and lymphatic system disorders) | 6 (6) | 0 (0) | 8 (8) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 6 (6) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Pyrexia (General disorders) | 3 (3) | 3 (5) | 8 (8) | 5 (6)
Bronchiolitis (Infections and infestations) | 1 (1) | 3 (7) | 3 (3) | 6 (6)
Candida nappy rash (Infections and infestations) | 1 (1) | 0 (0) | 9 (9) | 2 (5)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 4 (4)
Gastroenteritis (Infections and infestations) | 4 (5) | 2 (3) | 11 (11) | 8 (11)
Impetigo (Infections and infestations) | 2 (2) | 0 (0) | 2 (3) | 3 (3)
Lower respiratory tract infection (Infections and infestations) | 3 (4) | 0 (0) | 4 (5) | 2 (2)
Nasopharyngitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 3 (3)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 5 (6) | 5 (6)
Otitis media (Infections and infestations) | 4 (4) | 3 (11) | 7 (11) | 5 (6)
Otitis media acute (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 3 (5)
Pharyngitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 12 (26) | 4 (8) | 23 (47) | 22 (48)
Viral rash (Infections and infestations) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 11 (11) | 6 (8)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 3 (4) | 3 (3) | 2 (2)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 0 (0) | 6 (8) | 5 (5)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 9 (14) | 3 (3)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 4 (5) | 0 (0)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 6 (6) | 4 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 4 (4) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 8 (9) | 6 (7)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 4 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises on-going studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.